CLINICAL TRIAL: NCT04605874
Title: STUDY 3: A Multidisciplinary Examination of the Effects of Cigarillo Package Quantity on Consumption, Purchase Intentions, Risk Perceptions, Use and Exposure
Brief Title: Cigar Packaging Study
Acronym: CPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Strasser, Associate Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPCC 02021; 1U54CA229973 (NIH); 834476 (Other: IRB protocol number)
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Smoking
Keywords: Cigarillo, Behavior
MeSH Terms: conditions — Smoking; Behavior | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: This project will recruit current cigarillo users to a 20-day, randomized, parallel design protocol. After a 5-day period of smoking their own preferred brand of cigarillos, participants will begin a 15-day experimental period when they will be randomized to one of two conditions, 2 cigarillos per pack versus 4 cigarillos per pack, to examine how quantity per pack affects use patterns, including daily consumption and cigar smoking topography.
Who Masked: Participant
Masking Description: Participants will be informed that they will be supplied with study cigarillos, but will be unaware of their randomization condition, 2 cigarillos per pack versus 4 cigarillos per pack.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 cigarillos per pack (Experimental): After a 5-day period of smoking their own preferred brand of cigarillos, participants will begin a 15-day experimental period when they will be randomized to receive 2 cigarillos per pack.
  Interventions: Other: Package Quantity (cigarillos)
- 4 cigarillos per pack (Experimental): After a 5-day period of smoking their own preferred brand of cigarillos, participants will begin a 15-day experimental period when they will be randomized to receive 4 cigarillos per pack.
  Interventions: Other: Package Quantity (cigarillos)

INTERVENTIONS:
Other: Package Quantity (cigarillos) — After a 5-day period of smoking their own preferred brand of cigarillos, participants will begin a 15-day experimental period when they will be randomized to one of two conditions, 2 cigarillos per pack versus 4 cigarillos per pack.

SUMMARY:
The purpose of this study is to examine the effect of number of cigarillos per package on use behaviors, intensity of use and biomarkers of exposure.

DETAILED DESCRIPTION:
This laboratory-based study will aim to enroll 50 current cigarillo users to complete a 20-day, randomized, parallel design protocol. After a 5-day period of smoking their own preferred brand of cigarillos, participants will begin a 15-day experimental period when they will be randomized to one of two conditions, 2 cigarillos per pack versus 4 cigarillos per pack, to examine how quantity per pack affects use patterns, including daily consumption and cigar smoking topography. Participants will be asked to attend 2 in-person sessions on Days 5 and 20. On Days 0, 9, 12 and 16 participants will complete sessions with research staff remotely (i.e. by phone or video call). Sessions will occur every 3-5 days, for a total of 6 sessions across 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarillo smoker (i.e., smoked at least 50 cigarillos in their lifetime)
* Not currently undergoing smoking cessation treatment or planning to quit smoking over the duration of the study (~3 weeks).
* Plan to live in the area for the duration of the study.
* Willing to use study provided cigarillos.
* Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the combined Informed Consent and HIPAA form.
* Able to communicate fluently in English (i.e., speaking, writing, and reading).

Exclusion Criteria:

* Use of any nicotine-containing products other than cigarillos or cigarettes. Participants reporting isolated use of other nicotine containing products less than 5 times per month are eligible to participate.
* Current or impending enrollment in a smoking cessation program. Further, participants will be excluded for an attempt to quit smoking over the duration of the study period.
* History of substance abuse (other than nicotine dependence) in the past 12 months and/or currently receiving medical treatment for substance abuse. Attendance at alcoholics anonymous or narcotics anonymous meetings will not be considered medical treatment for the purposes of this protocol.
* Current alcohol consumption that exceeds 25 standard drinks/week.
* Women, including all individuals assigned as "female" at birth, who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period.
* Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the proper completion of the study procedures. Notable impairments will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Serious or unstable medical condition. Applicable conditions will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Lifetime history or current diagnosis of COPD, cardiovascular disease, or heart attack.
* Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.
* Current diagnosis of active major depression. Participants who maintain a diagnosis of major depression who have not experienced any major depressive episodes in the past 6 months and are stable on antidepressant medication(s) are eligible to participate.

Additional, general reasons for exclusion include:

* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
* Any circumstance, medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn for any of the aforementioned reasons at any point throughout the study.
* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Participants may be withdrawn at any point throughout the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Daily Cigarillo Consumption | Day 0 through Day 20
  Daily cigarillo consumption will be assessed by participant self-report throughout the 20-day study duration and verified through the collection of spent cigarillo "tips/ends" for all cigarillos smoked throughout the 15-day experimental period.
Smoking Topography | Day 5 through Day 20
  Topography data will be produced through a standardized video scoring procedure. Participants will video recorded to collect smoking topography data for all cigarillos smoked throughout the 15-day experimental period.
Total Nicotine Equivalents | Days 5 and 20
  Urine collected at Day 5 and Day 20 will be assessed for changes in total nicotine equivalents, nicotine plus its primary metabolites, across the experimental study period (Days 5-20). Total nicotine equivalents will be measured in nanograms per milliliter (ng per mL).
Total NNAL | Days 5 and 20
  Urine collected at Day 5 and Day 20 will be assessed for changes in NNAL, a biomarker of carcinogen exposure, across the experimental study period (Days 5-20). Total NNAL will be measured in nanograms per milliliter (ng per mL).

SECONDARY OUTCOMES:
Subjective Cigarillo Ratings (Visual Analog Scale [VAS] of Cigarillo Characteristics) | Day 5 through Day 20
  Participants will provide subjective ratings of each cigarillo smoked during each session using a 14-item, 100 mm visual analog scale (VAS) of cigarette characteristics. Anchors are item-specific (e.g., taste: 0 = "very bad," 100 = "very good"), with lower scores indicating less favorable ratings.
Cigarillo Craving (Questionnaire on Smoking Urges [QSU]) | Day 0 through Day 20
  Participants will report cigarillo craving at the onset of each session. Craving will be assessed using a summary score and two factor subscales (i.e., desire to smoke and craving due to anticipation of negative affect relief) from a 32-item Questionnaire on Smoking Urges (QSU). Participants will respond to each item along a 7-point scale (1=Strongly disagree; 7=Strongly agree).
Cigarillo Withdrawal (Withdrawal Symptom Checklist [WSC]) | Day 0 through Day 20
  Participants will report cigarillo withdrawal at the onset of each session. Withdrawal will be assessed using a summary score from the 20-item (21 items at Session 1 [Day 0]) revised version of the Withdrawal Symptom Checklist with a one-week frame of reference (WSC-W). Specifically, participants will respond regarding to how they felt in regards to each potential withdrawal symptom along a 4-point scale (0=Not Present; 3=Severe).
Cigar Evaluation (Cigar Evaluation Scale [CES]) | Day 5 through Day 20
  Participants will complete an 11-item questionnaire in regard to the cigarillo smoked during each session. Items on the questionnaire include subjective measures concerning taste, satisfaction, and physical effects.
Sensory Measure (Sensory Questionnaire [SQ]) | Day 5 through Day 20
  Participants will complete a 9-item questionnaire in regard to the cigarillo smoked during each session. Items on the questionnaire include subjective measures concerning puffs (e.g., satisfaction, perceived levels of nicotine, etc.) and puff sensations (i.e., how strong puffs were in a number of places such as the chest and nose).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research for Nicotine Addiction, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available to other researchers who contact the project Principal Investigator via email. Data will be available to such requests 1 year after the conclusion of recruitment.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year after the conclusion of recruitment.
Access Criteria: Researchers should contact the Principal Investigator via email.

DOCUMENTS (1):
  • Informed Consent Form (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04605874/ICF_000.pdf